CLINICAL TRIAL: NCT04543279
Title: Fostamatinib as a Single Agent or in Combination With Ruxolitinib for Treatment of Patients With Myelofibrosis With Severe Thrombocytopenia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Washington University School of Medicine (Other)
Collaborators: Rigel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202011080
Record Dates: First submitted 2020-09-08; First posted 2020-09-10 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Myelofibrosis; Thrombocytopenia
MeSH Terms: conditions — Primary Myelofibrosis; Thrombocytopenia | interventions — fostamatinib; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A: Fostamatinib (Experimental): The starting dose of fostamatinib is 100 mg twice daily (BID). After the first cycle, if no major dose related safety issue is observed and the platelet count is less than 50K/microL, then the fostamatinib dose will be increased to 150 mg BID for the next 2 cycles; otherwise the dose may be continued at 100 mg BID.
  Interventions: Drug: Fostamatinib
- Part B: Fostamatinib + Ruxolitinib (Experimental): After 3 cycles of fostamatinib monotherapy, all patients with a sustained platelet count ≥ 50K/microL, will continue on the current fostamatinib dose plus ruxolitinib at the recommended dose per standard prescribing guidelines for an additional 9 cycles.
  Patients who do not reach platelet count of at least 50K/microL but who achieve clinical benefit per the treating provider may continue on single agent fostamatinib for up to 12 total treatment cycles. If these patients achieve a sustained platelet count of ≥ 50K/microL at any point prior to Cycle 10 Day 1, then they may be eligible to enroll in Part B of the study and continue treatment with fostamatinib and ruxolitinib for the remainder of the study.
  Interventions: Drug: Fostamatinib; Drug: Ruxolitinib

INTERVENTIONS:
Drug: Fostamatinib — Fostamatinib will be supplied by Rigel Pharmaceuticals.
  Other Names: Tavalisse
Drug: Ruxolitinib — Ruxolitinib is commercially available.
  Other Names: Jakafi
  Arms: Part B: Fostamatinib + Ruxolitinib

SUMMARY:
Fostamatinib may improve thrombocytopenia in myelofibrosis patients with severe thrombocytopenia (platelet <50,000/microL) and allow them to initiate treatment with a JAK2 inhibitor, ruxolitinib. Additionally, fostamatinib monotherapy may also improve myelofibrosis related symptoms and splenomegaly.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of primary myelofibrosis or post-polycythemia vera/essential thrombocythemia myelofibrosis classified as high risk, intermediate-2 risk, or intermediate 1 risk by IPSS.
* Severe thrombocytopenia defined as platelet count < 50,000/microL (confirmed on at least two measurements over an 8-week period prior to start of study).
* At least 18 years of age.
* ECOG performance status ≤ 2
* Able to swallow pills
* Adequate bone marrow and organ function as defined below:

  * ANC ≥ 1000/microL
  * Peripheral blood blasts ≤ 10%
  * Albumin > 2.7 g/dL
  * Total bilirubin ≤ 1.5 x IULN; patients with Gilbert's syndrome may enroll if direct bilirubin ≤ 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 1.5 x IULN
  * Creatinine clearance > 30 mL/min by Cockcroft-Gault
* Female subjects must be either post-menopausal for at least 1 year or surgically sterile; or, if of childbearing potential, must not be pregnant or lactating and must agree to use a highly effective method of birth control throughout the duration of the trial and for 30 days following the last dose. Acceptable methods of birth control are defined as: hormonal contraception (pill, injection or implant) used consistently for at least 30 days prior to screening, an intrauterine device (IUD), or intrauterine hormone-releasing system (IUS), or true abstinence (i.e. abstinence is in line with the preferred and usual lifestyle of the subject.). Male subjects do not need to use contraception for fostamatinib because human studies showed minimal R406 in sperm.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* History of allogeneic stem cell transplant.
* Any solid tumor or hematologic malignancy (other than myelofibrosis) requiring active treatment at the time of study entry
* Currently receiving any other investigational agents.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to fostamatinib, ruxolitinib, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, or cardiac arrhythmia.
* Subject has uncontrolled or poorly controlled hypertension, defined as systolic blood pressure ≥130 mmHg or diastolic blood pressure ≥80 mmHg, whether or not the subject is receiving anti-hypertensive treatment.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry and prior to the first dose of fostamatinib.
* Known positive status for human immunodeficiency virus (HIV)
* Chronic, active, or acute viral hepatitis A, B, or C infection, or hepatitis B or C carrier.
* Treatment with strong CYP3A inhibitors or inducers within 14 days before the first dose of study drug. Strong CYP3A inhibitors and CYP3A inducers are not permitted during the study.
* Ongoing gastrointestinal medical condition such as Crohn's disease, inflammatory bowel disease, or chronic diarrhea that is not well controlled and could interfere with absorption of oral medication or be exacerbated by study medication
* Known hepatic cirrhosis or severe pre-existing hepatic impairment.
* Uncontrolled coagulopathy or bleeding disorder.
* Female patients who intend to donate eggs and male patients who intend to donate sperm during the course of this study or for 4 months after receiving the last dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Zhou, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Started | 3 | 0
Completed | 0 | 0
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: None of the participants in Part A received treatment on Part B.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 68 [66 to 79] |  | 68 [66 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 3 |  | 3
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Platelet Response (Part A)
Description: -Defined as an increase in platelet count ≥ 50K/microL with at least one more confirmatory platelet count separated by at least 2 weeks (in the absence of platelet transfusion) within the first 12 weeks of fostamatinib treatment
Time Frame: Week 12
Population: This outcome measure is only for Part A.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

2. Primary Outcome: Toxicity of Fostamatinib and Ruxolitinib Treatment (Part B)
Description: -Measured by number of adverse events, serious adverse events, and laboratory abnormalities
Time Frame: From start of treatment through 30 days after last day of study treatment (estimated to be approximately 40 weeks)
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants Eligible to Initiate Therapy With Ruxolitinib (Part A)
Time Frame: Through completion of fostamatinib treatment (12 weeks)
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

4. Secondary Outcome: Toxicity of Fostamatinib Treatment (Part A)
Description: -Measured by number of adverse events, serious adverse events, and laboratory abnormalities
Time Frame: From start of treatment through 30 days after last day of study treatment (estimated to be approximately 16 weeks)
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants
  Grade 3 neutrophil count decreased | 1 |
  Grade 3 white blood cell decreased | 1 |
  Grade 3 fatigue | 1 |
  Grade 1 chills | 2 |
  Grade 2 pain | 1 |
  Grade 1 fever | 1 |
  Grade 3 bacteremia | 1 |
  Grade 3 lung infection (pneumonia) | 1 |
  Grade 2 bruising | 1 |
  Grade 2 anorexia | 1 |
  Grade 3 joint pain secondary to arthritis | 1 |
  Grade 1 tendon cramps | 1 |
  Grade 3 neck pain | 1 |
  Grade 1 dyspnea | 1 |
  Grade 1 rash maculo-papular | 1 |
  Grade 2 hypertension | 1 |

5. Secondary Outcome: Number of Participants Who Permanently Discontinue Fostamatinib Due to Fostamatinib Related Adverse Events (Part A)
Time Frame: Through 12 weeks
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

6. Secondary Outcome: Number of Participants Who Require Treatment Interruption of Fostamatinib Due to Adverse Events (Part A)
Time Frame: Through 12 weeks
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 1 |

7. Secondary Outcome: Number of Participants Who Was Dose Escalated and Tolerated Fostamatinib Dose Greater Than 100 mg BID (Part A)
Time Frame: Through 12 weeks
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 2 |

8. Secondary Outcome: Number of Participants Who Achieve 35% or Greater Reduction in Spleen Volume as Determined by Ultrasound at Week 12 of Fostamatinib Treatment (Part A)
Time Frame: Week 12
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

9. Secondary Outcome: Change in Mean Spleen Volume as Determined by Ultrasound at Week 12 of Fostamatinib Treatment (Part A)
Time Frame: Week 12
Population: This outcome measure is for Part A only.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
cm^3 | 329.73 (169.04) |

10. Secondary Outcome: Number of Participants With 50% or Greater Improvement in Myeloproliferative Neoplasm - Symptom Assessment Form Total Symptom Score (Part A) From Baseline to Week 12
Description: -The Myeloproliferative Neoplasm - Symptom Assessment Form Total Symptom Score (MPN-SAF-TSS) has 10 questions for participants to rate their symptoms. The answers range from 0-absent to 10-worst imaginable. The total score for the questionnaire is 100. A higher score indicates worse symptoms.
Time Frame: Baseline and Week 12
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 1 |

11. Secondary Outcome: Number of Participants Who Achieve Platelet Transfusion Independence (Part A)
Time Frame: Through week 12
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

12. Secondary Outcome: Number of Participants With Anemia Who Achieve RBC Transfusion Independence (Part A)
Time Frame: Through week 12
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

13. Secondary Outcome: Number of Participants With Change in Marrow Fibrosis by WHO Grading (Part A)
Time Frame: Through week 12
Population: This outcome measure is for Part A only.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 3 | 0
Participants | 0 |

14. Secondary Outcome: Number of Participants With 35% or Greater Reduction in Spleen Volume as Determined by Ultrasound After 12 Weeks of Combination Treatment (Part B)
Time Frame: 12 weeks
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Number of Participants With 35% or Greater Reduction in Spleen Volume as Determined by Ultrasound After 12 Weeks of Combination Treatment (Part B)
Time Frame: At completion of combination treatment (estimated to be 36 weeks)
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Mean Reduction in Spleen Volume as Determined by Ultrasound After 12 Weeks of Combination Treatment (Part B)
Time Frame: 12 weeks
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Mean Reduction in Spleen Volume as Determined by Ultrasound After 12 Weeks of Combination Treatment (Part B)
Time Frame: At completion of combination treatment (estimated to be 36 weeks)
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Number of Participants With 50% or Greater Improvement in Total Symptom Score (Part B)
Time Frame: 12 weeks
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Number of Participants With 50% or Greater Improvement in Total Symptom Score (Part B)
Time Frame: At completion of combination treatment (estimated to be 36 weeks)
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Duration of Uninterrupted Ruxolitinib Treatment (Part B)
Time Frame: Up to 36 weeks
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Change in Marrow Fibrosis by WHO Grading (Part B)
Time Frame: At completion of combination treatment (estimated to be 36 weeks)
Population: No participants from Part A went on to receive treatment in Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from start of treatment through 30 days after last dose of treatment (median follow-up time 102 days, full range 89-145 days).
Description: No participants went on to receive Part B.
Arm/Group | Part A: Fostamatinib | Part B: Fostamatinib + Ruxolitinib
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Fostamatinib (N=3) | Part B: Fostamatinib + Ruxolitinib (N=0)
Lung infection (pneumonia) (Infections and infestations) | 1 | NA
Joint pain secondary to arthritis (Musculoskeletal and connective tissue disorders) | 1 | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Fostamatinib (N=3) | Part B: Fostamatinib + Ruxolitinib (N=0)
Chills (General disorders) | 2 | NA
Fatigue (General disorders) | 1 | NA
Fever (General disorders) | 1 | NA
Pain (General disorders) | 1 | NA
Bacteremia (Infections and infestations) | 1 | NA
Bruising (Injury, poisoning and procedural complications) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
White blood cell count decreased (Investigations) | 1 | NA
Anorexia (Metabolism and nutrition disorders) | 1 | NA
Tendon cramps (Musculoskeletal and connective tissue disorders) | 1 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | NA
Hypertension (Vascular disorders) | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT04543279/Prot_SAP_000.pdf